CLINICAL TRIAL: NCT01490034
Title: Effects of Learning and Food Form on Intake in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01DK079913-3; R01DK079913 (NIH)
Record Dates: First submitted 2011-12-05; First posted 2011-12-12 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
Keywords: obesity; energy intake; appetite; food form; beverage; learning; dietary compensation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Energy dense beverage (Experimental): Metabolic effects of consuming energy dense beverages before and after regular consumption
  Interventions: Behavioral: Metabolic effects of consuming energy dense beverages
- Energy dense solid food form (Experimental): Metabolic effects of consuming energy dense solid foods before and after regular exposure.
  Interventions: Behavioral: energy dense solid food
- Eenergy dilute beverages (Experimental): Metabolic effects of consumption of energy dilute beverages on a regular basis.
  Interventions: Behavioral: Energy dilute beverages
- Energy dilute solid food form (Experimental): Metabolic effects of consuming energy dilute sold foods before and after regular exposure.
  Interventions: Behavioral: Energy dilute solid food

INTERVENTIONS:
Behavioral: Metabolic effects of consuming energy dense beverages — Consumption of energy dense beverages for 2 weeks and monitoring physiological responses
  Arms: Energy dense beverage
Behavioral: energy dense solid food — Effects of consuming energy dense solid food for two weeks on physiological responses
  Arms: Energy dense solid food form
Behavioral: Energy dilute beverages — Effects of consuming energy dilute beverages for two weeks on physiological responses.
  Arms: Eenergy dilute beverages
Behavioral: Energy dilute solid food — Effects of consuming energy dilute solid food for two weeks on physiological responses
  Arms: Energy dilute solid food form

SUMMARY:
Due to the rising incidence of obesity, much emphasis has been placed on identifying mechanisms of increased energy intake. At this point, the mechanisms responsible for the recent increase in obesity prevalence have not been thoroughly examined. Pre-ingestive influences, such as cognitive factors, may play a larger role in creating an energy surplus than previously thought. Expectations about the satiating effect of a food may override the post-ingestive influences in dictating further consumption. In addition, obese individuals may exhibit a decreased compensatory response to foods as compared to lean individuals.

Understanding the effects of energy content, food form, and learning on satiation, satiety, and energy intake will allow for a greater understanding of the mechanisms of energy imbalance as a whole. Food choice is dictated by sensory properties and post-ingestive effects. By utilizing foods with similar sensory properties, the acquired knowledge derived from ingesting these foods can be monitored by analyzing subsequent intake at the same meal and at subsequent eating occurrences. It is hypothesized that the liquid food form will elicit weaker dietary compensation; that is, energy intake at other eating events will not be adjusted to compensate for that food. In addition, it is posited that the lower energy food will cause lower compensation postprandially. By having participants consume the same test food daily over a two week learning period, it is thought that they will show improved dietary compensation when the initial testing is repeated due to learned associations between food properties and metabolism.

DETAILED DESCRIPTION:
No expansion provided.

ELIGIBILITY:
Inclusion Criteria:

* Weight stable (<3 kg weight change within last 3 months)
* Constant habitual activity patterns (no deviation > 1x/wk at 30 min/session within last 3 months)
* Constant habitual diet patterns within last 3 months
* Willingness to eat a chocolate-flavored snack at test sessions and two week training period
* No allergies to any test foods
* Not planning to change use of medications known to influence appetite or metabolism
* Not diabetic
* No history of GI pathology
* Non-smoker for one year or more

Exclusion Criteria:

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
energy intake | 12 weeks
  Energy consumed over 12 weeks of intervention.
dietary compensation | 12 weeks
  spontaneous dietary adjustment in response to intervention
appetite | 12 weeks
  Effects of intervention on appetitive sensation such as hunger and fullness
effects of learning on energy intake | 12 weeks
  The effects of learning based on exposure to products that are high or low in energy and liquid or solid
Effects of food form on energy intake | 12 weeks
  The effects of food form on energy intake before and after chronic exposure to foods varying in food form and energy density
Effects of BMI on sensory learning | 12 weeks
  The effects of BMI on appetite, energy intake and dietary compensation

SECONDARY OUTCOMES:
Effects of personality traits on appetite, energy intake and compensation | 12 weeks
  Effects of personality traits related to feeding on appetite, energy intake and compensation following exposure to foods of different physical form, energy density and before and after learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Jones JB, Mattes RD. Effects of learning and food form on energy intake and appetitive responses. Physiol Behav. 2014 Oct;137:1-8. doi: 10.1016/j.physbeh.2014.06.016. Epub 2014 Jun 21. PMID 24955495